CLINICAL TRIAL: NCT01665417
Title: Randomized, Open Label, Positive Controlled, Multicenter Trial to Evaluate Icotinib as First-line and Maintenance Treatment in EGFR Mutated Patients With Lung Adenocarcinoma
Brief Title: Icotinib as First-line and Maintenance Treatment in EGFR Mutated Patients With Lung Adenocarcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV08
Record Dates: First submitted 2012-08-12; First posted 2012-08-15 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: EGFR Positive Non-small Cell Lung Cancer; Adenocarcinoma
Keywords: Icotinib; EGFR positive mutation; First-line treatment; Maintenance treatment
MeSH Terms: conditions — Adenocarcinoma | interventions — Drug Therapy; Pemetrexed; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Experimental Icotinib (Experimental): Icotinib: 125mg, oral administration, three times per day.
  Interventions: Drug: Experimental
- Chemotherapy Regimen 1 (Active Comparator): Chemotherapy Regimen 1：Pemetrexe 500 mg/m^2 on Day 1, Cisplatin 75 mg/m^2 on Day 1, 21 days/1 cycle, 2/4 cycles totally, until progression, withdrawal of consent, or unacceptable toxicity.
  Interventions: Drug: Chemotherapy
- Chemotherapy Regimen 2 (Active Comparator): Chemotherapy Regimen 2：Docetaxel 75 mg/m^2 on Day 1, Cisplatin 75 mg/m^2 on Day 1, 21 days/1 cycle, 2/4 cycles totally, until progression, withdrawal of consent, or unacceptable toxicity.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Experimental — Icotinib: 125mg, oral administration, three times per day.
  Other Names: BPI-2009; Commana
  Arms: Experimental Icotinib
Drug: Chemotherapy — Chemotherapy Regimen 1：Pemetrexe 500 mg/m^2 on Day 1, Cisplatin 75 mg/m^2 on Day 1, 21 days/1 cycle, 2/4 cycles totally, until progression, withdrawal of consent, or unacceptable toxicity.
  Other Names: Pemetrexe; ALIMTA
  Arms: Chemotherapy Regimen 1; Chemotherapy Regimen 2
Drug: Chemotherapy — Chemotherapy Regimen 2：Docetaxel 75 mg/m^2 on Day 1, Cisplatin 75 mg/m^2 on Day 1, 21 days/1 cycle, 2/4 cycles totally, until progression, withdrawal of consent, or unacceptable toxicity.
  Other Names: Docetaxel; Taxotere
  Arms: Chemotherapy Regimen 1; Chemotherapy Regimen 2

SUMMARY:
This study is designed to compare the efficacy and safety of first-line icotinib treatment and first-line chemotherapy followed by maintenance treatment with icotinib.

DETAILED DESCRIPTION:
This study is designed to compare the efficacy and safety of first-line icotinib treatment and first-line chemotherapy followed by maintenance with icotinib.

Primary endpoint:

Progression-free survival between first-line icotinib treatment and first-line chemotherapy followed by maintenance with icotinib

Secondary endpoint:

1. Overall survival between icotinib and chemotherapy
2. Time to Progression between icotinib and chemotherapy
3. Objective response rate and disease control rate between icotinib and chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of lung adenocarcinoma with measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded on CT); Patients must have previously untreated locally advanced or metastatic NSCLC; Patients must have lung cancer with a documented EGFR activating mutation (exon 19 deletion, L858R).

Exclusion Criteria:

* Prior chemotherapy Prior treatment with gefitinib, erlotinib, or other drugs that target EGFR Patients must not be receiving any other investigational agents Any evidence of interstitial lung disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-08; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 8 months
  PFS was defined as the time from the date of first dose of study medication to the date of first documentation of tumor progression or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival | 24 months
  OS was assessed via calculation of the time to death due to any cause from the date of randomization. A patient was censored at the last date they were known to be alive.
Time to Tumor Progression | 8 months
  TTP was defined as the time from the date of first dose of study medication to first documentation of objective tumor progression. If tumor progression data included more than 1 date, the first date was used. TTP (in weeks) was calculated as (first event date minus first dose date +1)/7. Kaplan-Meier method was used.
Objective response rate | 3 months
  Number of Subjects With Overall Confirmed Objective Disease Response According to the Response Evaluation Criteria in Solid Tumors(RECIST)1.1.
Number of participants with adverse events | 24 months
  Adverse events assessed by CTCAE4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jiao Shunchang, MD, Principal Investigator — Chinese People's Liberation Army (PLA) General Hospital; Fang Jian, MD, Study Director — Peking University Cancer Hospital & Institute; Bai Chunmei, MD, Study Director — Peking Union Medical College Hospital; Liu Wei, MD, Study Director — Hebei Provincal Tumor Hospital
Locations (1):
- Chinese People's Liberation Army (PLA) General Hospital, Beijing, Beijing Municipality, China